CLINICAL TRIAL: NCT04208334
Title: A Double-blind, Placebo-controlled Randomized Trial Phase II Evaluating the Effect of Curcumin for Treatment of Cancer Anorexia-Cachexia Syndrome in Patients With Stage III-IV of Head and Neck Cancer
Brief Title: The Effect of Curcumin for Treatment of Cancer Anorexia-Cachexia Syndrome in Patients With Stage III-IV of Head and Neck Cancer
Acronym: CurChexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R119h/61
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Cancer Cachexia; Head and Neck Cancer; Head and Neck Neoplasms
Keywords: Cancer cachexia; Head and neck cancer; Curcumin; Tumuric; Cancer anorexia cachexia
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental): Curcumin 4000mg/day x 60 days
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator): Placebo x 60 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — We give an Intervention arm to consume Curcumin 4000mg/day for 60 consecutive days.
  Arms: Curcumin
Other: Placebo — We give a control arm to consume placebo for 60 consecutive days.
  Arms: Placebo

SUMMARY:
A study of Curcumin to prevent cancer anorexia and cachexia Syndrom in locally advance and advance stage head and neck cancer (stage III, IV)

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer stage III-IV
* Cancer anorexia cachexia syndrome by 2011 Cancer cachexia an International Consensus
* Enteral feeding with Nasogastric Tube or Gastrostomy
* ECOG 0-2
* Normal Bone marrow, kidneys, and liver function
* Normal function of enteral digestion and absorption

Exclusion Criteria:

* Pregnancy
* History of allergy to Curcumin or herbal medicine
* History of Herbal medicine used
* History of Billiary of obstruction
* History of Antiplatelete or anticoagulant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 60 days after intervention
  We measure muscle mass by Bioelectrical Impedance Analysis (BIA)

SECONDARY OUTCOMES:
BMI | 60 days after intervention
  We measure BMI by Bioelectrical Impedance Analysis (BIA)
Hand grips muscle strength | 60 days after intervention
  We measure hand grips power by Hand grip test
serum NF-kB level | 60 days after intervention
  We measure serum NF-kB by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Tawasapon Thambamroong, MD, Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Argiles JM, Busquets S, Stemmler B, Lopez-Soriano FJ. Cancer cachexia: understanding the molecular basis. Nat Rev Cancer. 2014 Nov;14(11):754-62. doi: 10.1038/nrc3829. Epub 2014 Oct 9. PMID 25291291
- [Background] Puigserver P, Rhee J, Lin J, Wu Z, Yoon JC, Zhang CY, Krauss S, Mootha VK, Lowell BB, Spiegelman BM. Cytokine stimulation of energy expenditure through p38 MAP kinase activation of PPARgamma coactivator-1. Mol Cell. 2001 Nov;8(5):971-82. doi: 10.1016/s1097-2765(01)00390-2. PMID 11741533
- [Background] Meriggi F. Cancer Cachexia: One Step Ahead. Rev Recent Clin Trials. 2015;10(3):246-50. doi: 10.2174/1574887110666150916141351. PMID 26435290
- [Background] Argiles JM, Lopez-Soriano FJ. The ubiquitin-dependent proteolytic pathway in skeletal muscle: its role in pathological states. Trends Pharmacol Sci. 1996 Jun;17(6):223-6. doi: 10.1016/0165-6147(96)10021-3. PMID 8763200
- [Background] Glass DJ. Signaling pathways perturbing muscle mass. Curr Opin Clin Nutr Metab Care. 2010 May;13(3):225-9. doi: 10.1097/mco.0b013e32833862df. PMID 20397318
- [Background] Constantinou C, Fontes de Oliveira CC, Mintzopoulos D, Busquets S, He J, Kesarwani M, Mindrinos M, Rahme LG, Argiles JM, Tzika AA. Nuclear magnetic resonance in conjunction with functional genomics suggests mitochondrial dysfunction in a murine model of cancer cachexia. Int J Mol Med. 2011 Jan;27(1):15-24. doi: 10.3892/ijmm.2010.557. Epub 2010 Nov 10. PMID 21069263
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Result] Laviano A, Seelaender M, Sanchez-Lara K, Gioulbasanis I, Molfino A, Rossi Fanelli F. Beyond anorexia -cachexia. Nutrition and modulation of cancer patients' metabolism: supplementary, complementary or alternative anti-neoplastic therapy? Eur J Pharmacol. 2011 Sep;668 Suppl 1:S87-90. doi: 10.1016/j.ejphar.2011.06.060. Epub 2011 Jul 27. PMID 21810420
- [Result] Dewys WD, Begg C, Lavin PT, Band PR, Bennett JM, Bertino JR, Cohen MH, Douglass HO Jr, Engstrom PF, Ezdinli EZ, Horton J, Johnson GJ, Moertel CG, Oken MM, Perlia C, Rosenbaum C, Silverstein MN, Skeel RT, Sponzo RW, Tormey DC. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7. doi: 10.1016/s0149-2918(05)80001-3. PMID 7424938
- [Result] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Result] Evans WK, Makuch R, Clamon GH, Feld R, Weiner RS, Moran E, Blum R, Shepherd FA, Jeejeebhoy KN, DeWys WD. Limited impact of total parenteral nutrition on nutritional status during treatment for small cell lung cancer. Cancer Res. 1985 Jul;45(7):3347-53. PMID 2988769
- [Result] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Result] Cheng AL, Hsu CH, Lin JK, Hsu MM, Ho YF, Shen TS, Ko JY, Lin JT, Lin BR, Ming-Shiang W, Yu HS, Jee SH, Chen GS, Chen TM, Chen CA, Lai MK, Pu YS, Pan MH, Wang YJ, Tsai CC, Hsieh CY. Phase I clinical trial of curcumin, a chemopreventive agent, in patients with high-risk or pre-malignant lesions. Anticancer Res. 2001 Jul-Aug;21(4B):2895-900. PMID 11712783
- [Result] Dhillon N, Aggarwal BB, Newman RA, Wolff RA, Kunnumakkara AB, Abbruzzese JL, Ng CS, Badmaev V, Kurzrock R. Phase II trial of curcumin in patients with advanced pancreatic cancer. Clin Cancer Res. 2008 Jul 15;14(14):4491-9. doi: 10.1158/1078-0432.CCR-08-0024. PMID 18628464
- [Result] Thomas R, Williams M, Sharma H, Chaudry A, Bellamy P. A double-blind, placebo-controlled randomised trial evaluating the effect of a polyphenol-rich whole food supplement on PSA progression in men with prostate cancer--the U.K. NCRN Pomi-T study. Prostate Cancer Prostatic Dis. 2014 Jun;17(2):180-6. doi: 10.1038/pcan.2014.6. Epub 2014 Mar 11. PMID 24614693
- [Result] Srivastava DS, Dhaulakhandi DB. Role of NF-KB in Loss of Skeletal Muscle Mass in Cancer Cachexia and its Therapeutic Targets. AJCB. 2013;1(1):16.
- [Result] Thaloor D, Miller KJ, Gephart J, Mitchell PO, Pavlath GK. Systemic administration of the NF-kappaB inhibitor curcumin stimulates muscle regeneration after traumatic injury. Am J Physiol. 1999 Aug;277(2):C320-9. doi: 10.1152/ajpcell.1999.277.2.C320. PMID 10444409
- [Result] Gupta SC, Kim JH, Kannappan R, Reuter S, Dougherty PM, Aggarwal BB. Role of nuclear factor kappaB-mediated inflammatory pathways in cancer-related symptoms and their regulation by nutritional agents. Exp Biol Med (Maywood). 2011 Jun 1;236(6):658-71. doi: 10.1258/ebm.2011.011028. Epub 2011 May 12. PMID 21565893
- [Result] Panahi Y, Saadat A, Beiraghdar F, Sahebkar A. Adjuvant therapy with bioavailability-boosted curcuminoids suppresses systemic inflammation and improves quality of life in patients with solid tumors: a randomized double-blind placebo-controlled trial. Phytother Res. 2014 Oct;28(10):1461-7. doi: 10.1002/ptr.5149. Epub 2014 Mar 19. PMID 24648302
- [Result] Busquets S, Carbo N, Almendro V, Quiles MT, Lopez-Soriano FJ, Argiles JM. Curcumin, a natural product present in turmeric, decreases tumor growth but does not behave as an anticachectic compound in a rat model. Cancer Lett. 2001 Jun 10;167(1):33-8. doi: 10.1016/s0304-3835(01)00456-6. PMID 11323096
- [Result] Siddiqui RA, Hassan S, Harvey KA, Rasool T, Das T, Mukerji P, DeMichele S. Attenuation of proteolysis and muscle wasting by curcumin c3 complex in MAC16 colon tumour-bearing mice. Br J Nutr. 2009 Oct;102(7):967-75. doi: 10.1017/S0007114509345250. Epub 2009 Apr 27. PMID 19393114
- [Result] Gil da Costa RM, Aragao S, Moutinho M, Alvarado A, Carmo D, Casaca F, Silva S, Ribeiro J, Sousa H, Ferreira R, Nogueira-Ferreira R, Pires MJ, Colaco B, Medeiros R, Venancio C, Oliveira MM, Bastos MM, Lopes C, Oliveira PA. HPV16 induces a wasting syndrome in transgenic mice: Amelioration by dietary polyphenols via NF-kappaB inhibition. Life Sci. 2017 Jan 15;169:11-19. doi: 10.1016/j.lfs.2016.10.031. Epub 2016 Nov 22. PMID 27888116
- [Result] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Result] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Result] Reagan-Shaw S, Nihal M, Ahmad N. Dose translation from animal to human studies revisited. FASEB J. 2008 Mar;22(3):659-61. doi: 10.1096/fj.07-9574LSF. Epub 2007 Oct 17. PMID 17942826
- [Derived] Thambamroong T, Seetalarom K, Saichaemchan S, Pumsutas Y, Prasongsook N. Efficacy of Curcumin on Treating Cancer Anorexia-Cachexia Syndrome in Locally or Advanced Head and Neck Cancer: A Double-Blind, Placebo-Controlled Randomised Phase IIa Trial (CurChexia). J Nutr Metab. 2022 Jun 2;2022:5425619. doi: 10.1155/2022/5425619. eCollection 2022. PMID 35694030